CLINICAL TRIAL: NCT05407636
Title: A Randomized, Partially Masked, Controlled, Phase 3 Clinical Study to Evaluate the Efficacy and Safety of RGX-314 Gene Therapy in Participants With nAMD
Brief Title: Pivotal 2 Study of RGX-314 Gene Therapy in Participants With nAMD
Acronym: ASCENT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGX-314-3101; M23-409 (Other: AbbVie)
Record Dates: First submitted 2022-01-28; First posted 2022-06-07 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: AMD; nAMD; Wet Age-related Macular Degeneration; wAMD; WetAMD; CNV
Keywords: Age-Related Macular Degeneration; Neovascular Age-Related Macular Degeneration; Wet Macular Degeneration; Choroidal Neovascularization; Retinal Degeneration; Retinal Diseases; Eye Diseases; Ranibizumab; Aflibercept; Angiogenesis Inhibitors; Angiogenesis Modulating Agents; Growth Substances; Physiological Effects of Drugs; Growth Inhibitors; Antineoplastic Agents; Gene Therapy; Anti-vascular endothelial grown factory therapy; Anti-VEGF therapy; Macular Degeneration
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Choroidal Neovascularization; Retinal Degeneration; Retinal Diseases; Eye Diseases | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: 2 ABBV-RGX-314 treatment arms, 1 control arm (aflibercept)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: ABBV-RGX-314 administration is performed as an outpatient surgical procedure in an operating room, while the active control, aflibercept, is administered via intravitreal injection in an office setting. This study will be partially masked which will include masking of key study assessors and study drug dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABBV-RGX-314 Dose 1 (Experimental): ABBV-RGX-314 Dose 1 administered via subretinal delivery one time.
  Interventions: Genetic: ABBV-RGX-314 Dose 1
- ABBV-RGX-314 Dose 2 (Experimental): ABBV-RGX-314 Dose 2 administered via subretinal delivery one time.
  Interventions: Genetic: ABBV-RGX-314 Dose 2
- Control Arm (Active Comparator): Aflibercept administered via intravitreal injection approximately every 8 weeks
  Interventions: Biological: Aflibercept (EYLEA®)

INTERVENTIONS:
Genetic: ABBV-RGX-314 Dose 1 — AAV8 vector containing a transgene for anti-VEGF Fab (Dose 1)
  Other Names: RGX-314; surabgene lomparvovec
  Arms: ABBV-RGX-314 Dose 1
Genetic: ABBV-RGX-314 Dose 2 — AAV8 vector containing a transgene for anti-VEGF Fab (Dose 2)
  Other Names: RGX-314; surabgene lomparvovec
  Arms: ABBV-RGX-314 Dose 2
Biological: Aflibercept (EYLEA®) — 2.0 mg (0.05 mLsolution) administered by intravitreal injection approximately every 8 weeks after 3 monthly injections
  Other Names: Eylea (anti-VEGF agent)
  Arms: Control Arm

SUMMARY:
ABBV-RGX-314 (also known as RGX-314) is being developed as a novel one-time gene therapy for the treatment of neovascular (wet) age-related macular degeneration (wet AMD). Wet AMD is characterized by loss of vision due to new, leaky blood vessel formation in the retina. Wet AMD is a significant cause of vision loss in the United States, Europe and Japan, with up to 2 million people living with wet AMD in these geographies alone. Current anti-vascular endothelial growth factor (VEGF) therapies have significantly changed the landscape for treatment of wet AMD, becoming the standard of care due to their ability to prevent progression of vision loss in the majority of patients. These therapies, however, require life-long intraocular injections, typically repeated every four to 12 weeks in frequency, to maintain efficacy. Due to the burden of treatment, patients often experience a decline in vision with reduced frequency of treatment over time. ABBV-RGX-314 is being developed as a potential one-time treatment for wet AMD.

DETAILED DESCRIPTION:
This randomized, partially masked, controlled, Phase 3 clinical study will evaluate the efficacy and safety of ABBV-RGX-314 gene therapy in participants with nAMD. The study will evaluate 2 dose levels of RGX-314 gene therapy relative to an active comparator. The primary endpoint of this study is mean change in best-corrected visual acuity (BCVA) of ABBV-RGX-314 relative to aflibercept. Approximately 660 participants who meet the inclusion/exclusion criteria, will be enrolled into one of 3 arms.

A bilateral treatment substudy conducted at US sites is an open-label, partially randomized, parallel arm study to evaluate the safety and efficacy of subretinal ABBV-RGX-314 administered bilaterally in participants who have bilateral nAMD. Previously treated crossover participants from the control arm of the main study who crossed over and received ABBV-RGX-314 in the study eye will receive the same ABBV-RGX-314 dose in the contralateral eye (ie, same dose as in the study eye), and newcomers (participants who have not been randomized in an ABBV-RGX-314 study) and untreated crossover participants (ongoing control participants in the main study who have completed Week 54 but have not crossed over to receive ABBV-RGX-314 in the main study) will be randomized in a 2:1 ratio to receive ABBV-RGX-314 Dose 1 or ABBV-RGX-314 Dose 2 in both eyes. Up to 15 participants who qualify for the substudy will be enrolled and followed for a minimum of 50 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years and ≤ 89 years
2. An ETDRS BCVA letter score between ≤ 78 and ≥ 40 in the study eye
3. Diagnosis of subfoveal choroidal neovascularization (CNV) secondary to AMD in the study eye previously treated with anti-VEGF
4. Must be pseudophakic (at least 12 weeks postcataract surgery) in the study eye
5. Willing and able to provide written, signed informed consent for this study
6. Participants must have demonstrated a meaningful response to anti-VEGF therapy at study entry

Inclusion Criteria (Bilateral Treatment Substudy)*:

1. An ETDRS BCVA letter score between ≤ 83 and ≥ 40 in both eyes
2. Diagnosis of subfoveal choroidal neovascularization (CNV) secondary to AMD in both eyes
3. Must be pseudophakic (at least 12 weeks postcataract surgery) in both eyes
4. Willing and able to provide written, signed informed consent for this study
5. Newcomers must have active disease in the study eye; crossover participants must have active disease in the eye not treated in the main study

Exclusion Criteria:

1. CNV or macular edema in the study eye secondary to any causes other than AMD
2. Subfoveal fibrosis or atrophy in the study eye
3. Any condition in the investigator's opinion that could limit VA improvement in the study eye
4. Active or history of retinal detachment, or current retinal tear that cannot be treated, in the study eye
5. Advanced glaucoma or history of secondary glaucoma in the study eye
6. Myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 6 months
7. History of intraocular surgery in the study eye within 12 weeks prior to randomization
8. History of intravitreal therapy in the study eye, such as intravitreal steroid injection or investigational product, other than anti-VEGF therapy, in the 6 months prior to Screening Visit 1
9. Prior treatment with gene therapy

Exclusion Criteria (Bilateral Treatment Substudy)*:

1. CNV or macular edema in either eye secondary to any causes other than AMD
2. Subfoveal fibrosis or atrophy in either eye
3. Any condition in the investigator's opinion that could limit VA improvement in either eye
4. Active or history of retinal detachment, or current retinal tear that cannot be treated in either eye
5. Advanced glaucoma or history of secondary glaucoma in either eye
6. Myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 6 months
7. History of intraocular surgery in either eye within 12 weeks prior to randomization
8. History of intravitreal therapy in either eye, such as intravitreal steroid injection or investigational product, other than anti-VEGF therapy, in the 6 months prior to screening
9. Prior treatment with gene therapy (*) For previously treated crossover participants, criteria apply to the eye not treated in the main study only.

Note: Other inclusion/exclusion criteria apply

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Best Corrected Visual Acuity (BCVA) | At Week 54
  BCVA measured by Early Treatment Diabetic Retinopathy Study (ETDRS)
Bilateral Treatment Substudy: Incidence of ocular AEs and any SAEs | Week 50
  AEs and SAEs through Week 50

SECONDARY OUTCOMES:
Proportion of participants with ≤ 2 supplemental anti-VEGF injections | Through Week 54 (ABBV-RGX-314 randomized participants only)
  Proportion of supplemental anti-VEGF injections
Proportion of participants with no supplemental anti-VEGF injections | Through Week 54 (ABBV-RGX-314 randomized participants only)
  Proportion of supplemental anti-VEGF injections
Incidences of ocular and overall SAEs over 54 weeks | Through Week 54
  AEs over 54 weeks
Proportion of participants with worsened BCVA | Week 54
  Proportion with worsened BCVA
Proportion of participants with improved BCVA | Week 54
  Proportion with improved BCVA
Proportion of participants (1) gaining or losing greater than 0 letters; (2) maintaining vision compared with baseline as per BCVA | Week 54
  Proportion gaining or losing greater than 0 letters based on ETDRS score; proportion maintaining vision
Mean change from baseline in BCVA for participants who received 0 or more supplemental anti-VEGF injection (ABBV-RGX-314 randomized participants) | Week 54
  Mean change in BCVA based on ETDRS score for participants who received 0 or more supplemental anti-VEGF injection
Mean change from Week 54 to Week 108 in BCVA (control arm participants who cross over to ABBV-RGX-314) | Week 54 to Week 108
  Mean change in BCVA based on ETDRS score
Mean change from baseline in central retinal thickness (CRT) as measured by SD-OCT | Week 54
  Mean change in CRT as measured by SD-OCT
Mean change from Week 54 to Week 108 in CRT as measured by SD-OCT (control arm participants who cross over to ABBV-RGX-314) | Week 54 to Week 108
  Mean change in CRT as measured by SD-OCT
Mean change from baseline in center point thickness (CPT) as measured by SD-OCT | Week 54
  Mean change in CPT as measured by SD-OCT
Mean change from Week 54 to Week 108 in CPT, as measured by SD-OCT (control arm participants who cross over to ABBV-RGX-314) | Week 54 to Week 108
  Mean change in CPT as measured by SD-OCT
Proportion of participants with a reduction in anti-VEGF injection annualized rate | Through Week 54
  Proportion of participants with a reduction in anti-VEGF injection annualized rate compared with the prior year
Supplemental anti-VEGF injection annualized rate in the ABBV-RGX-314 arms | Through Week 54
  Supplemental anti-VEGF injection annualized rate
Percent reduction in anti-VEGF injection annualized rate after Week 58 through Week 108 relative to the year prior to the study (control arm participants who cross over to ABBV-RGX 314) | After Week 58 to Week 108
  Percent reduction in anti-VEGF injection annualized rate
Supplemental anti-VEGF injection annualized rate after Week 58 through Week 108 (control arm participants who cross over to ABBV-RGX-314) | After Week 58 through Week 108
  Supplemental anti-VEGF injection annualized rate
Time to first supplemental anti-VEGF injection after the Week 2 injection (ABBV-RGX-314 randomized participants) | Through Week 54
  Time to first supplemental anti-VEGF injection
Time to first supplemental anti-VEGF injection after the Week 58 injection in the control arm participants who cross over to ABBV-RGX-314 | After Week 58 through Week 108
  Time to first supplemental anti-VEGF injection
Mean change from baseline in NEI VFQ-25 (composite score) | Week 54 and Week 108
  Mean change in NEI VFQ-25 (composite score) at Week 54 and (control arm participants who cross over to ABBV-RGX-314) Week 108
Mean change from baseline in MacTSQ (composite score) | Week 54 and Week 108
  Mean change from baseline in MacTSQ (composite score) at week 54 and (control arm participants who cross over to ABBV-RGX-314) at Week 108
Aqueous ABBV-RGX-314 transgene product (TP) concentration (ABBV-RGX-314 randomized participants) | Week -2, Week 14, Week 38, and Week 54
  Aqueous ABBV-RGX-314 TP concentration
Aqueous ABBV-RGX-314 TP concentration (control arm participants who cross over to ABBV-RGX-314) | Week 54, Week 74, Week 90, and Week 108
  Aqueous ABBV-RGX-314 TP concentration
Serum ABBV-RGX-314 TP concentrations (at select sites) | Week -2, Week 14, Week 38, and Week 54
  Serum ABBV-RGX-314 TP concentration
Immunogenicity measurements (ABBV-RGX-314 randomized participants) | Week -2, Week 14, Week 38, and Week 54
  Immunogenicity measurements (serum antibodies to AAV8 and serum antibodies to ABBV-RGX-314 TP)
Immunogenicity measurements (control arm participants who cross over to ABBV-RGX-314) | Week 54, Week 74, Week 90, and Week 108
  Immunogenicity measurements (serum antibodies to AAV8 and serum antibodies to ABBV-RGX-314 TP)
Bilateral Treatment Substudy: Incidence of nonocular AEs and any AEs of special interest | Week 50
  Nonocular AEs and AEs of Special Interest
Bilateral Treatment Substudy: Mean change from Baseline in BCVA at assessed time points | Through Week 50
  BCVA measured by ETDRS
Bilateral Treatment Substudy: Mean change from Baseline in CRT at assessed time points | Through Week 50
  Mean change in CRT as measured by SD-OCT
Bilateral Treatment Substudy: Supplemental anti-VEGF injection annualized rate | Through Week 50
  Supplemental anti-VEGF injection annualized rate
Bilateral Treatment Substudy: Mean number of supplemental anti-VEGF injections | Through Week 50
  Mean supplemental anti-VEGF injections
Bilateral Treatment Substudy: Proportion of participants with no supplemental anti-VEGF injections | Through Week 50
  Proportion of participants with no supplemental anti-VEGF injections
Bilateral Treatment Substudy: Proportion of participants with ≤ 2 supplemental anti-VEGF injections | Through Week 50
  Proportion of participants with ≤ 2 supplemental anti-VEGF injections
Bilateral Treatment Substudy: Aqueous humor and serum ABBV-RGX-314 TP concentrations | Week 26, Week 34, Week 50
  Aqueous humor and serum ABBV-RGX-314 TP concentrations
Bilateral Treatment Substudy: Immunogenicity measurements (serum anti-ABBV-RGX-314 TP antibodies, serum antiAAV8 antibodies) and enzyme-linked immunospot at assessed time points | Week 18, Week 34, Week 50
  Immunogenicity measurements

CONTACTS AND LOCATIONS:
Locations (181):
- United States (107):
  - Barnet Dulaney Eye Center-Phoenix /ID# 256340, Phoenix, Arizona
  - Retinal Research Institute /ID# 256238, Phoenix, Arizona
  - Retina Macula Institute of Arizona /ID# 271026, Scottsdale, Arizona
  - California Retina Consultants - Bakersfield /ID# 256240, Bakersfield, California
  - Retina Vitreous Assoc Med Grp /ID# 256246, Beverly Hills, California
  - Retinal Diagnostic Center /ID# 256262, Campbell, California
  - The Retina Partners - Encino /ID# 259660, Encino, California
  - Retina Consultants of Orange County /ID# 256267, Fullerton, California
  - Hamilton Glaucoma Center Shiley Eye Center UCSD /ID# 256320, La Jolla, California
  - California Retina Consultants - Oxnard - North Ventura Road /ID# 262883, Oxnard, California
  - Byers Eye Institute Stanford /ID# 262853, Palo Alto, California
  - Retina Consultants of San Diego /ID# 256258, Poway, California
  - Kaiser Permanente - Riverside Medical Center /ID# 262413, Riverside, California
  - University of California Davis Health /ID# 256317, Sacramento, California
  - Retinal Consultants Medical Group, Inc. - Greenback /ID# 256353, Sacramento, California
  - Orange County Retina Medical Group /ID# 256286, Santa Ana, California
  - Macula Retina Vitreous Center - Torrance /ID# 270247, Torrance, California
  - Bay Area Retina Associates - Walnut Creek - Lennon Lane /ID# 268513, Walnut Creek, California
  - Retina Consultants of Southern Colorado /ID# 256285, Colorado Springs, Colorado
  - Southwest Retina Research Center /ID# 256261, Durango, Colorado
  - Colorado Retina Associates /ID# 256378, Lakewood, Colorado
  - Eye Care Center of Northern Colorado-Longmont /ID# 256380, Longmont, Colorado
  - Retina Consultants, P.C. /ID# 273610, Manchester, Connecticut
  - Duplicate_Rand Eye Institute /ID# 256337, Deerfield Beach, Florida
  - National Ophthalmic Research Institute /ID# 256344, Fort Myers, Florida
  - Vitreoretinal Associates, P.A. /ID# 256266, Gainesville, Florida
  - Florida Retina Consultants /ID# 256321, Lakeland, Florida
  - Florida Retina Institute - Orlando /ID# 256373, Orlando, Florida
  - Retina Specialty Institute /ID# 256268, Pensacola, Florida
  - Fort Lauderdale Eye Institute /ID# 266011, Plantation, Florida
  - Retina Vitreous Associates of Florida - St. Petersburg /ID# 256279, St. Petersburg, Florida
  - Center for Retina and Macular Disease /ID# 256335, Winter Haven, Florida
  - Georgia Retina - Marietta /ID# 256264, Marietta, Georgia
  - Retina Consultants of Hawaii /ID# 256278, ‘Aiea, Hawaii
  - Illinois Retina Associates-Oak Park Office /ID# 256375, Chicago, Illinois
  - Northwestern Medicine Fertility and Reproductive Medicine /ID# 256379, Chicago, Illinois
  - University Retina and Macula Associates /ID# 256288, Lemont, Illinois
  - University Retina and Macula Associates /ID# 256287, Oak Forest, Illinois
  - Springfield Clinic /ID# 256371, Springfield, Illinois
  - Retina Partners Midwest, PC /ID# 256277, Indianapolis, Indiana
  - John-Kenyon American Eye Institute -New Albany /ID# 256283, New Albany, Indiana
  - Wolfe Eye Clinic - West Des Moines /ID# 256314, West Des Moines, Iowa
  - Retina Associates - Lenexa /ID# 258296, Lenexa, Kansas
  - Maine Eye Center - Marginal Way Campus /ID# 256391, Portland, Maine
  - Greater Baltimore Medical Ctr /ID# 256392, Baltimore, Maryland
  - Johns Hopkins Hospital /ID# 256236, Baltimore, Maryland
  - Mid Atlantic Retina Specialists - Hagerstown /ID# 256310, Hagerstown, Maryland
  - MA Eye & Ear Infirmary /ID# 262430, Boston, Massachusetts
  - Ophthalmic Consultants of Boston /ID# 256233, Boston, Massachusetts
  - Vitreo Retinal Associates - Worcester /ID# 266008, Worcester, Massachusetts
  - Retina Associates of Michigan /ID# 256393, Grand Blanc, Michigan
  - Associated Retinal Consultants /ID# 256269, Royal Oak, Michigan
  - VitreoRetinal Surgery PLLC DBA Retina Consultants of Minnesota /ID# 256272, Edina, Minnesota
  - Mayo Clinic - Rochester /ID# 258295, Rochester, Minnesota
  - Mississippi Retina Associates /ID# 270934, Madison, Mississippi
  - Midwest Vision Research Foundation at Pepose Vision Institute /ID# 258993, Chesterfield, Missouri
  - University of Missouri Hospital /ID# 262474, Columbia, Missouri
  - Washington University School of Medicine - St. Louis /ID# 256383, St Louis, Missouri
  - Sierra Eye Associates /ID# 256239, Reno, Nevada
  - Envision Ocular, LLC /ID# 256367, Bloomfield, New Jersey
  - Monmouth Retina Consultants /ID# 275895, Little Silver, New Jersey
  - Columbia University of New York - Edward S. Harkness Eye Institute /ID# 256342, New York, New York
  - Retina Associates of Western New York /ID# 256374, Rochester, New York
  - Western Carolina Retinal Associates /ID# 256355, Asheville, North Carolina
  - Duke Eye Center /ID# 256245, Durham, North Carolina
  - Graystone Eye /ID# 256424, Hickory, North Carolina
  - Cincinnati Eye Institute /ID# 256247, Blue Ash, Ohio
  - Retina Associates of Cleveland-Middleburg Heights /ID# 256280, Cleveland, Ohio
  - Cleveland Clinic - Cleveland /ID# 256282, Cleveland, Ohio
  - Ohio State University /ID# 256275, Columbus, Ohio
  - Midwest Retina /ID# 276644, Dublin, Ohio
  - Retina Vitreous Center, Research /ID# 256284, Edmond, Oklahoma
  - University of Pennsylvania /ID# 258995, Philadelphia, Pennsylvania
  - Mid Atlantic Retina /ID# 256232, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center /ID# 258994, Pittsburgh, Pennsylvania
  - Charleston Neuroscience Institute - Beaufort /ID# 256385, Beaufort, South Carolina
  - Charleston Neurosciences Institute /ID# 256336, Charleston, South Carolina
  - Charleston Neurosciences Institute /ID# 256351, Charleston, South Carolina
  - Palmetto Retina Center-Florence /ID# 256244, Florence, South Carolina
  - Black Hills Regional Eye Institute /ID# 262872, Rapid City, South Dakota
  - Southeastern Retina Associates - Chattanooga /ID# 258992, Chattanooga, Tennessee
  - Charles Retina Institute /ID# 256237, Germantown, Tennessee
  - Southeastern Retina Associates - Johnson City /ID# 256396, Johnson City, Tennessee
  - Tennessee Retina - Nashville /ID# 256388, Nashville, Tennessee
  - Vanderbilt University Medical Center /ID# 256372, Nashville, Tennessee
  - Retina Research Institute of Texas /ID# 256263, Abilene, Texas
  - Austin Research Center for Retina /ID# 256265, Austin, Texas
  - Austin Clinical Research, LLC /ID# 256274, Austin, Texas
  - Retina Consultants of Texas - Bellaire /ID# 256377, Bellaire, Texas
  - Star Retina - Burleson /ID# 256376, Burleson, Texas
  - Ophthalmology Surgery Center of Dallas /ID# 256259, Dallas, Texas
  - Texas Retina Associates - Fort Worth /ID# 256326, Fort Worth, Texas
  - Austin Retina Associates - Round Rock /ID# 256387, Round Rock, Texas
  - RCTX - San Antonio Retina Center /ID# 259661, San Antonio, Texas
  - Stone Oak Surgery Center /ID# 256381, San Antonio, Texas
  - Brown Retina Institute /ID# 256382, San Antonio, Texas
  - Retina Center Of Texas (Rct) - Southlake /ID# 256281, Southlake, Texas
  - Rocky Mountain Retina Consultants /ID# 256369, Murray, Utah
  - Retina Associates of Utah /ID# 256276, Salt Lake City, Utah
  - Piedmont Eye Center /ID# 256386, Lynchburg, Virginia
  - Wagner Macula & Retina Center - Norfolk /ID# 256260, Norfolk, Virginia
  - Retina Institute of Virginia /ID# 256394, Richmond, Virginia
  - Vistar Eye Center /ID# 271024, Roanoke, Virginia
  - Pacific Northwest Retina /ID# 258999, Bellevue, Washington
  - Retina Center NW, PLLC /ID# 256395, Silverdale, Washington
  - Spokane Eye Clinic /ID# 256338, Spokane, Washington
  - Gundersen Health System - La Crosse Medical Center /ID# 276012, La Crosse, Wisconsin
- Canada (10):
  - Calgary Retina Consultants /ID# 258997, Calgary, Alberta
  - Alberta Retina Consultants /ID# 265599, Edmonton, Alberta
  - Retina Surgical Associates /ID# 270958, New Westminster, British Columbia
  - University of British Columbia - Eye Care Centre, Vancouver General Hospital /ID# 266014, Vancouver, British Columbia
  - Vitreous Retina Macula Specialists of Toronto /ID# 258299, Etobicoke, Ontario
  - Ottawa Hospital Research Institute /ID# 258998, Ottawa, Ontario
  - Retina Centre of Ottawa /ID# 259659, Ottawa, Ontario
  - Toronto Retina Institute /ID# 265602, Toronto, Ontario
  - Sunnybrook Health Sciences Centre /ID# 270690, Toronto, Ontario
  - Duplicate_CHU de Quebec-Universite Laval /ID# 258996, Québec, Quebec
- France (10):
  - Centre Hospitalier Universitaire de Nice - Hôpital Pasteur /ID# 262418, Nice, Alpes-Maritimes
  - Hôpital de la Croix Rousse - Groupement Hospitalier Nord /ID# 262409, Lyon, Auvergne-Rhône-Alpes
  - CHU Dijon /ID# 262410, Dijon, Cote-d Or
  - Chu De Toulouse - Hopital Pierre Paul Ricquet /ID# 262411, Toulouse, Occitanie
  - Hopitaux Universitaires Paris Centre-Hopital Cochin /ID# 262415, Paris, Paris
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 262408, Nantes, Pays de la Loire Region
  - Clinique Juge /ID# 262417, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hosp Intercommunal de Creteil /ID# 262407, Créteil, Val-de-Marne
  - Clinique Honoré Cave /ID# 262225, Montauban
  - AP-HP - Groupe Hospitalier 10e - Hopital Lariboisiere /ID# 262406, Paris
- Germany (7):
  - Universitaetsklinikum Freiburg /ID# 262495, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 262494, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Bonn /ID# 262498, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Muenster /ID# 262499, Münster, North Rhine-Westphalia
  - Klinikum Ludwigshafen /ID# 262497, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 262493, Hamburg
  - Knappschaftsklinikum Saar /ID# 262496, Püttlingen
- Hungary (3):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 262646, Debrecen, Hajdú-Bihar
  - Budapest Retina Intezet /ID# 262647, Budapest
  - Ganglion Orvosi Központ /ID# 264550, Pécs
- Italy (10):
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale S.Anna /ID# 262896, Cona, Ferrara
  - IRCCS Ospedale San Raffaele /ID# 263035, Milan, Milano
  - ASST Fatebenefratelli Sacco /ID# 263273, Milan, Milano
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 264074, Naples, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 263037, Rome, Roma
  - IRCCS Fondazione G.B. Bietti per lo studio e la ricerca in Oftalmologia- ONLUS /ID# 262897, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 263536, Negrar, Verona
  - A.O.U. Consorziale Policlinico di Bari /ID# 262500, Bari
  - ASL 2 Abruzzo Lanciano-Vasto-Chieti /ID# 263923, Chieti
  - ASU FC - P.O. Universitario Santa Maria della Misericordia /ID# 263036, Udine
- Japan (9):
  - Nagoya University Hospital /ID# 267350, Nagoya, Aichi-ken
  - Fukushima Medical University Hospital /ID# 258411, Fukushima, Fukushima
  - Kobe City Eye Hospital /ID# 256948, Kobe, Hyōgo
  - Hyogo Medical University Hospital /ID# 257893, Nishinomiya-shi, Hyōgo
  - Kagoshima University Hospital /ID# 257053, Kagoshima, Kagoshima-ken
  - Kyoto University Hospital /ID# 267351, Kyoto, Kyoto
  - University of Miyazaki Hospital /ID# 262879, Miyazaki, Miyazaki
  - Shiga University of Medical Science /ID# 266862, Ōtsu, Shiga
  - Juntendo University Hospital /ID# 258715, Bunkyo-ku, Tokyo
- Emanuelli Research & Development Center LLC /ID# 256231, Arecibo, Puerto Rico
- Spain (10):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 262632, Santiago de Compostela, A Coruna
  - Hospital Universitari de Bellvitge /ID# 262641, L'Hospitalet de Llobregat, Barcelona
  - Hospital Arruzafa /ID# 262634, Córdoba, Cordoba
  - Complejo Hospitalario Universitario Insular-Materno Infantil de Gran Canaria /ID# 262633, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 262635, Majadahonda, Madrid
  - Institut Clínic d'Oftalmologia (ICOF). Hospital Clínic d'Oftalmologia. /ID# 262644, Barcelona
  - Instituto de Microcirugía Ocular /ID# 262642, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 262637, Barcelona
  - Hospital Universitario 12 de Octubre /ID# 262636, Madrid
  - Clinica Baviera /ID# 270146, Madrid
- United Kingdom (14):
  - Stoke Mandeville Hospital /ID# 277343, Aylesbury, Buckinghamshire
  - Hammersmith Hospital /ID# 271621, London, England
  - Gloucestershire Royal Hospital /ID# 277362, Gloucester, Gloucestershire
  - Moorfields Eye Hospital /ID# 263038, London, Greater London
  - The Retina Clinic London /ID# 262304, London, Greater London
  - University Hospital Southampton NHS Foundation Trust /ID# 262307, Southampton, Hampshire
  - Oxford University Hospitals NHS Foundation Trust /ID# 262306, Oxford, Oxfordshire
  - Leeds Teaching Hospitals NHS Trust /ID# 277366, Leeds, West Yorkshire
  - Bradford Royal Infirmary /ID# 273164, Bradford
  - Bristol Eye Hospital /ID# 271619, Bristol
  - Liverpool University Hospitals NHS Foundation Trust /ID# 262305, Liverpool
  - Manchester University NHS Foundation Trust /ID# 262404, Manchester
  - Royal Victoria Infirmary /ID# 277368, Newcastle upon Tyne
  - Sunderland Eye Infirmary /ID# 271620, Sunderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=RGX-314-3101